CLINICAL TRIAL: NCT06449456
Title: A Comparison of Exercise Capacity, Muscle Functions, Physical Fitness, and Physical Activity Levels in Children With Congenital Adrenal Hyperplasia and Healthy Controls
Brief Title: Exercise Capacity, Physical Fitness, and Physical Activity Levels in Children With CAH
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Professor, Hacettepe University
Other Study IDs: SBA 24/096
Record Dates: First submitted 2024-05-27; First posted 2024-06-10 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Congenital Adrenal Hyperplasia; Exercise Capacity; Physical Activity; Quality of Life
Keywords: Congenital Adrenal Hyperplesia; Physical Fitness; Exercise Capacity; Physical Activity; Quality of Life; Heart Rate Variability - HRV
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Congenital Adrenal Hyperplasia: Patients between the ages of 8-18 years who have been diagnosed with Congenital Adrenal Hyperplasia
- Healthy Controls: Age and sex matched healthy controls between the ages of 8-18 years

SUMMARY:
Congenital Adrenal Hyperplesia (CAH) is a group of automosal recessive disorders that develop due to a deficiency of one of the five enyzmes necessary for cortisol synthesis in the adrenal cortex. Research indicates a predisposition in children and adolescents with CAH towards adverse metabolic changes such as obesity, hypertension, insulin resistance and increased intima-media thickness. This study aims to compare the extent to which children and adolescents with CAH are effected in terms of respiratory and peripheral muscle strength, exercise capasity, physical fitness and physical activity levels compared o their matched healthy individuals.

DETAILED DESCRIPTION:
Congenital adrenal hyperplasia (CAH) is a group of autosomal recessive diseases caused by the deficiency of one of the five enzymes necessary for cortisol synthesis in the adrenal cortex. Dysfunction in cortisol synthesis, as seen in other enzyme deficiencies, leads to an increase in adrenocorticotropic hormone (ACTH) secretion, resulting in hypertension and hypokalemia. Additionally, patients with CAH exhibit excess androgens alongside cortisol deficiency. İn CAH treatment, glucocorticoids are used to suppress androgen production in the adrenal cortex. Deficiency in glucocorticoids and mineralocorticoids, as well as excess androgens, can contribute to the development of adverse metabolic and cardiovascular anomalies.

Ongoing research has revealed a predisposition for adverse metabolic changes in children and adolescents with CAH, including obesity, hypertension, insulin resistance, and increased intima-media thickness, which can increase the risk of developing cardiovascular disease in adulthood. Furthermore, subclinical left ventricular diastolic dysfunction has been observed in adolescents with CAH. İn these patients, due to the deficiency of epinephrine there is an increased tendency for hypoglycemia under stress conditions.

These metabolic changes can lead to impaired exercise performance in patients with CAH, consequently affecting their quality of life.

A study involving twenty classic CAH adolescents and twenty healthy counterparts demonstrated that classic CAH patients exhibited reduced exercise capacity with lower peak workload and higher peak systolic blood pressure during exercise. However, there is a lack of research in the literature comparing respiratory and peripheral muscle strength, daily life activities, physical fitness, and levels of physical activity in children and adolescents with CAH to their healthy peers.

ELIGIBILITY:
Inclusion Criteria for CAH Group:

* Diagnosed with Congenital Adrenal Hyperplasia
* Aged between 8-18 years
* Providing voluntary consent from both themselves and their parents
* Able to cooperate

Exclusion Criteria for CAH Groups:

- Having any systemic disease that may affect the measurement parameters

Inclusion Criteria for Healthy Group:

* Not having any chronic diseases
* Aged between 8-18 years
* Willing to participate in the study
* Able to cooperate

Exclusion Criteria for Healthy Group:

* Not willing to participate in the study
* Presence of cooperation and communication problems

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents aged 8-18 years diagnosed with classical congenital adrenal hyperplasia (CAH) who apply to and are followed up by the Hacettepe University Hospital, Pediatric Endocrinology Department will be accepted for the study. The snowball sampling method will be used for our control group. The investigators plan to contact the patient's relatives and then contact someone else in the same way.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Respiratory Muscle Strength | 1 day
  Respiratory muscle strength will be measured using a portable, electronic mouth pressure measurement device (Micro Medical MicroMPM, UK). The best of three measurements for Maximal inspiratory pressure (MIP) and Maximal expiratory pressure (MEP) will be selected. Real MIP and MEP values and the percentages of expected values based on age and gender will be used in the analyses.
Peripheral Muscle Strength | 1 day
  Peripheral muscles'strength will be assessed using the K-Force hand dynamometer.
Physical Fitness Level | 1 day
  It will be evaluated with the Fitnessgram test battery.
Functional Exercise Capacity | 1 day
  It will be measured using the 6-Minute Walk Test.
Physical Activity Level | 1 day
  The Physical Activity Level will be assessed using the Physical Activity Questionnaire for Adolescents (PAQ-A) and the Physical Activity Questionnaire for Children (PAQ-C). The scores for PAQ-A and PAQ-C range from 9 to 45, with higher scores indicating better physical activity levels. The results of both questionnaires will be presented separately. The PAQ-A score will be reported as a distinct outcome measure for adolescents, and the PAQ-C score will be reported as a distinct Outcome Measure for children. This approach ensures a clear evaluation of physical activity levels in both age groups.
Handgrip strength | 1 day
  Jamar hand dynamometer (Jamar®, California, USA) will be used to measure grip strength.

SECONDARY OUTCOMES:
Anthropometric Measurements | 1 day
  Anthropometric measurements will include separate measurements of waist and hip circumference, and calculations of the waist/hip ratio and waist/height ratio.
Body composition | 1 day
  Body composition will be evaluated using bioelectric impedance analysis (Body Composition Analyzer MC-780MA). Measurements will include fat mass, fat-free mass, and water percentage. Each of these measurements will be reported as separate outcome measures. Fat mass will be reported in kilograms, fat-free mass in kilograms, and water percentage as a percentage of total body weight.
Participation | 1 day
  Quality of life will be assessed using the Pediatric Outcome Data Collection Instrument (PODCI) child and adolescent form. Scores for all dimensions range from 0 to 100, with 100 indicating the highest level of function or participation.
Heart Rate Variability | 1 day
  HRV will be assessed by measuring it with the Polar H10 device before, after, and during the recovery phase of the 6-minute walk test, specifically in the first and second minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru CALIK KUTUKCU, PhD, Principal Investigator — Ankara, Hacettepe University, Türkiye, 06100 Contact: Phd 0903123051576 Ext.195 ecalik85@gmail.com
Locations (1):
- Hacettepe University, Ankara, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No